CLINICAL TRIAL: NCT01890187
Title: Repeatability and Reproducibility of Cirrus HD-OCT Measurements of Illumination Areas Under the Retinal Pigment Epithelium
Status: Completed | Type: Observational
Sponsor: Carl Zeiss Meditec, Inc. (Industry)
Collaborators: DataMed Devices Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HD-OCT-GA-2010-2
Record Dates: First submitted 2013-06-24; First posted 2013-07-01 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Advanced Dry AMD With Geographic Atrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Advanced dry AMD with geographic atrophy: Patients diagnosed with advanced dry AMD with geographic atrophy

SUMMARY:
The objective of this study is to determine the repeatability and reproducibility of the Cirrus HD-OCT measurement of illumination areas under the retinal pigment epithelium (RPE).

DETAILED DESCRIPTION:
This is a prospective, single site study. Ocular history and examination will be conducted on consented subjects to determine further participation in the study. The study will be divided into two phases. In Phase 1, the inter-device variability of Cirrus HD-OCT measurements of illumination areas under the RPE will be determined. In Phase 2, the inter-operator variability of Cirrus HD-OCT measurements of illumination areas under the RPE will be determined. In each of these phases, the Macular Cube 200 x 200 scan and the Macular Cube 512 x 128 scan will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 50 years of age and older diagnosed to have advanced dry AMD with geographic atrophy.
* Geographic atrophy lesions should:

  * Not be greater than 5 mm at the widest diameter. The entire lesion(s) should fit into the 6x6 mm scan area of the Cirrus HD-OCT.
  * Not be smaller than 1.25 mm2.
  * Not be confluent with peri-papillary atrophy.
  * Not be combined with other lesions such as CNV.
* Able and willing to make the required study visits.
* Able and willing to give consent and follow study instructions.

Exclusion Criteria:

* History of retinal surgery, laser photocoagulation, and/or radiation therapy to the eye.
* Evidence of other retinal diseases of the eye, including wet AMD, diabetic retinopathy, diabetic macular edema, or significant vitreomacular traction.
* Thick media opacity or inability to fixate that precludes obtaining acceptable scans.
* Concomitant use of hydrochloroquine or chloroquine.
* Unable to make the required study visits.
* Unable to give consent or follow study instructions.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2010-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Coefficient of variation for area of increased illumination under the RPE (mm^2) | Single visit observation

SECONDARY OUTCOMES:
Coefficient of variation of the closest distance to fovea | Single visit observation

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Lujan, MD, Principal Investigator — West Coast Retina
Locations (1):
- West Coast Retina, Walnut Creek, California, United States